CLINICAL TRIAL: NCT06000371
Title: Cutoff Value of Ankle Brachial Pressure Index for Vacuum Assisted Closure Application in Diabetic Foot Ulcers
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: MS.20.03.1083
Record Dates: First submitted 2023-07-31; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Vacuum assisted Closure application — Vacuum assisted Closure Application in Diabetic Foot Ulcers

SUMMARY:
Abstract Objective To verify cutoff value of ankle brachial pressure index at which diabetic foot ulcers get benefit from vacuum assisted closure application and to assess impact of its application on ankle brachial pressure index value in the presence of peripheral arterial disease.

Methods An observational descriptive prospective analytic study had been performed.56 patients were enrolled in the study. All patients had three sessions of vacuum-assisted closure application. Debridement was done when indicated. Ulcer dimensions were measured before and after each session, while ankle brachial pressure index was measured before the first session .

DETAILED DESCRIPTION:
Introduction Diabetes Mellitus (DM) is a chronic disease, which is considered a global public health problem that leads to major clinical, economic, social, and quality of patient life issues (1). 15% of diabetics will develop a diabetic foot ulcer (DFU) during their lifetime, which is an exceedingly expensive and disabling complication of diabetes mellitus. (2).

Assessment of foot perfusion is a crucial step in treatment of patients with DFU. The ankle-brachial pressure index (ABPI) is a simple, quick, non-invasive tool (3). The key elements of effective DFU management are clinical awareness, appropriate blood glucose levels, regular foot exams, therapeutic footwear that fits the patient, off-loading, local wound care, and the identification and treatment of osteomyelitis and ischemia (4).

Multiple adjuvant therapies have been studied to decrease DFU healing times and amputation rates. These therapies include negative pressure wound therapy (vacuum-assisted closure), non-surgical debridement agents, oxygen therapies, human growth factors, energy based therapies, and systemic therapies(5).Cellular and/ or tissue based product (CTPs) may result in higher average number of ulcer free months and lower average number of amputations and resections compared to standard of care (SOC) alone (6).

Negative pressure wound therapy (NPWT) is a non-invasive therapy that removes fluid from wounds, prepares the wound bed for closure, reduces edema, and promotes the creation and perfusion of granulation tissue by applying regulated negative pressure using a vacuum-assisted closure (VAC) device (7). NPWT is indicated in traumatic, acute wounds, sub-acute wounds (i.e. dehisced incisions), chronic open wounds (stasis ulcers and diabetic ulcers), pressure ulcers, flaps and meshed graft (8).

We conducted this this study to verify cutoff value of ABPI at which diabetic foot ulcers get benefit from VAC application.

Methods A single-center prospective observational study had been performed. Between March 2020 and May 2021, 56 patients with DFUs underwent VAC application in the Department of Vascular Surgery. The inclusion criteria consisted of the following: the patient ≥40 years with unhealed diabetic foot ulcers belonged to grade 1 or grade 2 (in both wound and infection categories of wound, ischemia and wound infection " WIFI classification) . Patients with immunocompromised status, varicose veins, chronic venous insuffiency, foot ulcers belonged to grade 3 (in both wound and infection categories of WIFI classification) . All patients who were involved in the study gave their written consent.

The patients were subjected to history taking including history of foot ulceration, amputation, symptoms of claudication, neurologic changes, vascular surgery and medical comorbidities. The site, shape, base and margins of the ulcer had been clinically examined. The clinical manifestations of infection including erythema, warmth, swelling, pain or tenderness were searched for. Proper neurological and vascular examination had been applied to all included feet. The following investigations were done: duplex U/S on arterial system (for all patients), X-ray (in case of suspected infected collections or osteomyelitis) and CT angiography (when duplex is inconclusive).

Procedure description:

Prior to VAC application, ABPI was measured and documented with using of Bistos hi dop vascular Doppler with 8MHZ probe (Bistos Co., Ltd. Galmachi-ro, Jungwon-gu, Seongnam-si, Gyeonggi-do, Korea) and mercurial sphygmomanometer (ALPK2, 300v velcro cuff, Japan) according to the procedure described by the American College of Cardiology (ACC) and the American Heart Association (AHA) guidelines (9) and ulcer was prepared by debridement of devitalized tissue, proper hemostasis and wound irrigation with saline .

Then, length, width and depth of the ulcer were measured by metal ruler and documented. The ulcer was gently filled with foam, ensuring that the foam was slightly above the ulcer edge. The drain was placed between foam layers. The drape was sized and trimmed to cover the entire ulcer as well as about 3-5 cm of intact skin around it. The drape shouldn't be stretched or under tension. Adhesive plaster was used at edges to maintain sealing and negative suction .

The dressing drain was attached to canister tube with opening the clamp. The suction pressure was adjusted at-120 mmHg with intermittent mode. If the patient experienced bleeding despite good hemostasis or pain that was not relieved by analgesics, pressure can be reduced by 10mmHg. Power button was pressed to turn on Smith& Nephew Renesys EZ plus NPWT device (Smith & Nephew Medical Ltd. Hull HU3 2BN, England. The patient was informed about steps of disconnection and maximum period of disconnection 2hours /day. Patient or his/her relative was informed about causes of alarm e.g. low pressure, full canister, line blockage and low battery and how to manage them.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥40 years.
* Unhealed diabetic foot ulcers.
* Ulcers belonged to grade 1 or grade 2 (in both wound and infection categories "WIFI" classification) .

Exclusion Criteria:

* Immunocompromised patients.
* Patient with varicose veins and chronic venous insufficiency.
* Foot ulcers belonged to grade 3 (in both wound and infection categories of WIFI classification)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient ≥40 years with unhealed diabetic foot ulcers belonged to grade 1 or grade 2 (in both wound and infection categories of WIFI classification) .
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
Dimensions of diabetic foot ulcer (manual measurement of length, width and depth of the ulcer by metal ruler). | Up to3 weeks
  Change of dimensions of diabetic foot ulcers. The higher values mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mansoura university, Principal Investigator — MU
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Bonoto BC, de Araújo VE, Godói IP, de Lemos LLP, Godman B, Bennie M, et al. Efficacy of mobile apps to support the care of patients with diabetes mellitus: a systematic review and meta-analysis of randomized controlled trials. JMIR mHealth and uHealth. 2017;5(3):e4. 2. Yazdanpanah L, Nasiri M, Adarvishi S. Literature review on the management of diabetic foot ulcer. World journal of diabetes. 2015;6(1):37. 3. Hajibandeh S, Hajibandeh S, Shah S, Child E, Antoniou GA, Torella F. Prognostic significance of ankle brachial pressure index: a systematic review and meta-analysis. Vascular. 2017;25(2):208-24. 4. Mavrogenis AF, Megaloikonomos PD, Antoniadou T, Igoumenou VG, Panagopoulos GN, Dimopoulos L, et al. Current concepts for the evaluation and management of diabetic foot ulcers. EFORT open reviews. 2018;3(9):513-25. 5. Everett E, Mathioudakis N. Update on management of diabetic foot ulcers. Annals of the New York Academy of Sciences. 2018;1411(1):153. 6. Serena TE, Yaakov RA, Mostow EN. Use of Cellular and Tissue-based Product in the Treatment of Diabetic Foot Ulcers. The Journal of Foot and Ankle Surgery (Asia-Pacific). 2016;3(2):92-6. 7. Lone AM, Zaroo MI, Laway BA, Pala NA, Bashir SA, Rasool A. Vacuum-assisted closure versus conventional dressings in the management of diabetic foot ulcers: a prospective case-control study. Diabetic foot & ankle. 2014;5(1):23345. 8. Yadav S, Rawal G, Baxi M. Vacuum assisted closure technique: a short review. The Pan African Medical Journal. 2017;28. 9. Aboyans V, Criqui MH, Abraham P, Allison MA, Creager MA, Diehm C, et al. Measurement and interpretation of the ankle-brachial index: a scientific statement from the American Heart Association. Circulation. 2012;126(24):2890-909.